CLINICAL TRIAL: NCT01785849
Title: A Randomized, Double-blind, Placebo-controlled, Phase 3 Study to Assess the Efficacy and Safety of AMG 416 in the Treatment of Secondary Hyperparathyroidism in Subjects With Chronic Kidney Disease on Hemodialysis
Brief Title: Efficacy and Safety of Etelcalcetide (AMG 416) in the Treatment of Secondary Hyperparathyroidism (SHPT) in Patients With Chronic Kidney Disease on Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20120229; KAI-4169-006 (Other: KAI Pharmaceuticals, Inc (wholly owned subsidiary of Amgen Inc.)); 2012-002805-23 (EudraCT Number)
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Hyperparathyroidism, Secondary
Keywords: Secondary Hyperparathyroidism (SHPT), chronic kidney disease (CKD), hemodialysis, parathyroid hormone (PTH), hypocalcemia, bone and mineral metabolism
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic; Hypocalcemia | interventions — etelcalcetide hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Etelcalcetide (Experimental): Participants received etelcalcetide administered by intravenous bolus injection at the end of each hemodialysis session three times a week, for 26 weeks.
  Interventions: Drug: Etelcalcetide
- Placebo (Placebo Comparator): Participants received placebo administered by intravenous bolus injection at the end of each hemodialysis session, three times per week (TIW) for 26 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etelcalcetide — Administered intravenously three times per week. The starting dose was 5 mg. The dose may have been increased at 4-week intervals by 2.5 mg or 5 mg on the basis of the predialysis parathyroid hormone and corrected calcium concentrations obtained in the prior week. The minimum dose was 2.5 mg and the maximum dose was 15 mg.
  Other Names: AMG 416; KAI-4169
  Arms: Etelcalcetide
Drug: Placebo — Administered intravenously (IV) three times per week.
  Arms: Placebo

SUMMARY:
This study is designed to assess the efficacy and safety of etelcalcetide compared with placebo in the treatment of SHPT in patients with chronic kidney disease (CKD) receiving hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Subject understands the study procedures and agrees to participate in the study by giving written informed consent.
* Subject is 18 years of age or older.
* Subject must be receiving hemodialysis 3 times weekly for at least 3 months
* Subject agrees to not participate in another study of an investigational agent during the study.
* Other Inclusion Criteria may apply

Exclusion Criteria:

* Currently receiving treatment in another investigational device or drug study, or ended treatment on another investigational device or drug study(s) within 8 weeks prior to screening.
* Other investigational procedures while participating in this study are excluded.
* Anticipated or scheduled parathyroidectomy during the study period.
* Subject has received a parathyroidectomy within 3 months prior to dosing.
* Anticipated or scheduled kidney transplant during the study period.
* Subject has known sensitivity to any of the products or components to be administered during dosing.
* Subject has participated in a prior clinical trial of AMG 416 (also referred to as KAI-4169).
* Subject has received cinacalcet within the 4 weeks prior to screening labs (treatment with cinacalcet is prohibited during the study).
* Subject has an unstable medical condition based on medical history, physical examination, and routine laboratory tests, or is otherwise unstable in the judgment of the Investigator.
* Other Exclusion Criteria may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2013-03-12 (Actual); Primary Completion 2014-05-22 (Actual); Study Completion 2014-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (105):
- United States (47):
  - Research Site, Birmingham, Alabama
  - Research Site, Pine Bluff, Arkansas
  - Research Site, Azusa, California
  - Research Site, Covina, California
  - Research Site, Lakewood, California
  - Research Site, Los Angeles, California
  - Research Site, Lynwood, California
  - Research Site, Northridge, California
  - Research Site, Ontario, California
  - Research Site, Panorama City, California
  - Research Site, Sacramento, California
  - Research Site, Whittier, California
  - Research Site, Pembroke Pines, Florida
  - Research Site, Meridian, Idaho
  - Research Site, Evanston, Illinois
  - Research Site, Springfield, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Pontiac, Michigan
  - Research Site, Southgate, Michigan
  - Research Site, Tupelo, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, Reno, Nevada
  - Research Site, Amherst, New York
  - Research Site, Brooklyn, New York
  - Research Site, Rosedale, New York
  - Research Site, The Bronx, New York
  - Research Site, Yonkers, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Allentown, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Orangeburg, South Carolina
  - Research Site, Sumter, South Carolina
  - Research Site, Columbia, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Grand Prairie, Texas
  - Research Site, Houston, Texas
  - Research Site, Mansfield, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Tyler, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Mechanicsville, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Bluefield, West Virginia
- Australia (4):
  - Research Site, Liverpool, New South Wales
  - Research Site, St Leonards, New South Wales
  - Research Site, Parkville, Victoria
  - Research Site, Prahan, Victoria
- Austria (3):
  - Research Site, Graz
  - Research Site, Linz
  - Research Site, Vienna
- Belgium (5):
  - Research Site, Aalst
  - Research Site, Baudour
  - Research Site, Brussels
  - Research Site, Leuven
  - Research Site, Liège
- Canada (4):
  - Research Site, Brampton, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Czechia (5):
  - Research Site, Hradec Králové
  - Research Site, Prague
  - Research Site, Praha 4 - Nusle
  - Research Site, Slavkov u Brna
  - Research Site, Třinec
- France (5):
  - Research Site, Nantes
  - Research Site, Poitiers
  - Research Site, Reims
  - Research Site, Saint-Ouen
  - Research Site, Salouël
- Germany (4):
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Kiel
  - Research Site, Villingen-Schwenningen
- Hungary (5):
  - Research Site, Baja
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Kaposvár
  - Research Site, Pécs
- Israel (3):
  - Research Site, Ashkelon
  - Research Site, Nahariya
  - Research Site, Tel Aviv
- Italy (5):
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Pavia
  - Research Site, San Fermo Della Battaglia (CO)
  - Research Site, Verona
- Poland (4):
  - Research Site, Bialystok
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Zamość
- Research Site, Saint Petersburg, Russia
- Spain (3):
  - Research Site, Santander, Cantabria
  - Research Site, Barcelona, Catalonia
  - Research Site, Madrid
- United Kingdom (7):
  - Research Site, Cambridge
  - Research Site, Coventry
  - Research Site, Glasgow
  - Research Site, London
  - Research Site, Nottingham
  - Research Site, Salford
  - Research Site, Sheffield

REFERENCES:
- [Background] Block GA, Bushinsky DA, Cunningham J, Drueke TB, Ketteler M, Kewalramani R, Martin KJ, Mix TC, Moe SM, Patel UD, Silver J, Spiegel DM, Sterling L, Walsh L, Chertow GM. Effect of Etelcalcetide vs Placebo on Serum Parathyroid Hormone in Patients Receiving Hemodialysis With Secondary Hyperparathyroidism: Two Randomized Clinical Trials. JAMA. 2017 Jan 10;317(2):146-155. doi: 10.1001/jama.2016.19456. PMID 28097355
- [Background] Kroenke MA, Weeraratne DK, Deng H, Sloey B, Subramanian R, Wu B, Serenko M, Hock MB. Clinical immunogenicity of the d-amino acid peptide therapeutic etelcalcetide: Method development challenges and anti-drug antibody clinical impact assessments. J Immunol Methods. 2017 Jun;445:37-44. doi: 10.1016/j.jim.2017.03.005. Epub 2017 Mar 6. PMID 28274835
- [Background] Stollenwerk B, Iannazzo S, Akehurst R, Adena M, Briggs A, Dehmel B, Parfrey P, Belozeroff V. A Decision-Analytic Model to Assess the Cost-Effectiveness of Etelcalcetide vs. Cinacalcet. Pharmacoeconomics. 2018 May;36(5):603-612. doi: 10.1007/s40273-017-0605-2. PMID 29392552
- [Background] Stollenwerk B, Iannazzo S, Cooper K, Belozeroff V. Exploring the potential value of improved care for secondary hyperparathyroidism with a novel calcimimetic therapy. J Med Econ. 2017 Oct;20(10):1110-1115. doi: 10.1080/13696998.2017.1360309. Epub 2017 Aug 14. PMID 28803497
- [Background] Chen P, Narayanan A, Wu B, Gisleskog PO, Gibbs JP, Chow AT, Melhem M. Population Pharmacokinetic and Pharmacodynamic Modeling of Etelcalcetide in Patients with Chronic Kidney Disease and Secondary Hyperparathyroidism Receiving Hemodialysis. Clin Pharmacokinet. 2018 Jan;57(1):71-85. doi: 10.1007/s40262-017-0550-4. PMID 28508378
- [Background] Block GA, Chertow GM, Sullivan JT, Deng H, Mather O, Tomlin H, Serenko M. An integrated analysis of safety and tolerability of etelcalcetide in patients receiving hemodialysis with secondary hyperparathyroidism. PLoS One. 2019 Mar 15;14(3):e0213774. doi: 10.1371/journal.pone.0213774. eCollection 2019. PMID 30875390
- [Background] Cunningham J, Block GA, Chertow GM, Cooper K, Evenepoel P, Iles J, Sun Y, Urena-Torres P, Bushinsky DA. Etelcalcetide Is Effective at All Levels of Severity of Secondary Hyperparathyroidism in Hemodialysis Patients. Kidney Int Rep. 2019 Apr 16;4(7):987-994. doi: 10.1016/j.ekir.2019.04.010. eCollection 2019 Jul. PMID 31317120
- [Background] Wolf M, Block GA, Chertow GM, Cooper K, Fouqueray B, Moe SM, Sun Y, Tomlin H, Vervloet M, Oberbauer R. Effects of etelcalcetide on fibroblast growth factor 23 in patients with secondary hyperparathyroidism receiving hemodialysis. Clin Kidney J. 2019 Apr 26;13(1):75-84. doi: 10.1093/ckj/sfz034. eCollection 2020 Feb. PMID 32082556
- [Background] Hain D, Tomlin H, Gibson C. Administration of Etelcalcetide for the Treatment of Secondary Hyperparathyroidism in Patients with CKD-MBD on Hemodialysis: A Nephrology Nursing Perspective. Nephrol Nurs J. 2019 May-Jun;46(3):315-290. PMID 31199098
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 111 centers in the US, Canada, Europe, Israel, Russian Federation, and Australia. The first participant was enrolled on 12 March 2013 and the last participant enrolled on 08 November 2013.
Pre-assignment Details: Eligible participants were randomized in a 1:1 ratio to etelcalcetide or placebo. Randomization was stratified by mean screening parathyroid hormone (PTH) (< 600 pg/mL, 600 to ≤ 1000 pg/mL, and > 1000 pg/mL), prior cinacalcet use and region (North America or non-North America).
Groups:
- Etelcalcetide: Participants received etelcalcetide administered by intravenous bolus injection at the end of each hemodialysis session, TIW, for 26 weeks. The starting dose was 5 mg and may have been increased at weeks 5, 9, 13 and 17 to achieve a predialysis PTH ≤ 300 pg/mL.
Period: Overall Study
Arm/Group | Placebo | Etelcalcetide
Started | 254 | 254
Received Treatment | 254 | 251
Completed | 193 | 220
Not Completed | 61 | 34
Not completed — Death | 7 | 9
Not completed — Protocol Specified Criteria | 29 | 1
Not completed — Withdrawal by Subject | 15 | 12
Not completed — Sponsor Decision | 0 | 1
Not completed — Lost to Follow-up | 10 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Etelcalcetide | Total
Number analyzed (Participants) | 254 | 254 | 508
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (14.5) | 58.4 (14.6) | 57.7 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 103 | 217
  Male | 140 | 151 | 291
Race [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 5 | 8
  Black (or African American) | 69 | 72 | 141
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  White | 175 | 173 | 348
  Other | 4 | 4 | 8
  Missing | 1 | 0 | 1
Stratification Factor: Mean Screening Serum Parathyroid Hormone (PTH) [Number; unit: participants] — Mean screening parathyroid hormone (PTH) obtained within 2 weeks prior to randomization.
  participants
    < 600 pg/mL | 84 | 87 | 171
    ≥ 600 to ≤ 1000 pg/mL | 114 | 115 | 229
    > 1000 pg/mL | 56 | 52 | 108
Stratification Factor: Cinacalcet Use Within 8 Weeks of Randomization [Number; unit: participants]
  Yes | 34 | 33 | 67
  No | 220 | 221 | 441
Stratification Factor: Region [Number; unit: participants]
  North America | 129 | 132 | 261
  Non-North America | 125 | 122 | 247
Parathyroid Hormone (PTH) [Mean (Standard Deviation); unit: pg/mL] | 819.7 (386.0) | 848.7 (520.4) | 834.2 (457.9)
Phosphorus [Mean (Standard Deviation); unit: mg/dL] — Data were available for 250 subjects in each treatment group.
  mg/dL | 5.78 (1.60) | 5.95 (1.59) | 5.87 (1.59)
Corrected Calcium [Mean (Standard Deviation); unit: mg/dL] | 9.61 (0.60) | 9.65 (0.66) | 9.63 (0.63)
Corrected Calcium Phosphorus Product (cCa x P) [Mean (Standard Deviation); unit: mg²/dL²] — Data were available for 249 and 250 subjects in each treatment group respectively.
  mg²/dL² | 55.54 (15.81) | 57.37 (15.51) | 56.46 (15.67)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a > 30% Decrease From Baseline in Mean PTH During the Efficacy Assessment Phase
Description: Participants who did not have any scheduled assessments during the EAP were considered non-responders.
Time Frame: Baseline and the efficacy assessment phase (EAP; defined as Weeks 20 to 27, inclusive).
Population: The full analysis set, consisting of all randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 254 | 254
percentage of participants | 8.3 | 74.0
Statistical Analysis 1: Comparison: Placebo vs Etelcalcetide; A Cochran-Mantel-Haenszel test stratified by screening PTH category (< 600, ≥ 600 to ≤ 1000, and > 1000 pg/mL), recent cinacalcet use within 8 weeks before randomization (yes and no), and region (North America and non-North America) was used to compare the primary endpoint of proportion of participants with > 30% reduction from baseline in PTH during the EAP between etelcalcetide and placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 32.46, 95% CI 2-sided [18.71 to 56.31]

2. Secondary Outcome: Percentage of Participants With Mean Predialysis Parathyroid Hormone ≤ 300 pg/mL During the Efficacy Assessment Phase
Description: Participants who had no scheduled assessments during the EAP were considered non-responders.
Time Frame: Baseline and the efficacy assessment phase (Week 20 to Week 27)
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 254 | 254
percentage of participants | 5.1 | 49.6
Statistical Analysis 1: Comparison: Placebo vs Etelcalcetide; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by screening PTH category, recent cinacalcet use within 8 weeks before randomization, and region; Odds Ratio (OR) = 22.08, 95% CI 2-sided [11.47 to 42.48]

3. Secondary Outcome: Percent Change From Baseline in Predialysis PTH During the Efficacy Assessment Phase
Time Frame: Baseline and the Efficacy Assessment Phase (Week 20 to Week 27)
Population: Full analysis set participants with observed data
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 219 | 229
percent change | 13.00 (2.81) | -55.11 (1.94)
Statistical Analysis 1: Comparison: Placebo vs Etelcalcetide; Test type: Superiority or Other; p < 0.001, Repeated Measures Mixed Effects Model; Repeated measures mixed-effects model included treatment, stratification factors, visit, and treatment by visit interaction as covariates; Mean Difference = -71.11, 95% CI 2-sided [-77.77 to -64.46], Standard Error of Mean 3.39 — Etelcalcetide - Placebo

4. Secondary Outcome: Percent Change From Baseline in Predialysis Corrected Calcium During the Efficacy Assessment Phase
Time Frame: Baseline and the efficacy assessment phase (Week 20 to Week 27)
Population: Full analysis set participants with observed data
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 219 | 229
percent change | 1.18 (0.29) | -7.29 (0.53)
Statistical Analysis 1: Comparison: Placebo vs Etelcalcetide; Test type: Superiority or Other; p < 0.001, Repeated Measures Mixed Effects Model; [statistical method as in outcome 3, analysis 1]; Mean Difference = -8.38, 95% CI 2-sided [-9.52 to -7.23], Standard Error of Mean 0.58 — Etelcalcetide - Placebo

5. Secondary Outcome: Percent Change From Baseline in Predialysis Corrected Calcium Phosphorus Product During the Efficacy Assessment Phase
Time Frame: Baseline and the efficacy assessment phase (Week 20 to Week 27)
Population: Full analysis set participants with observed data
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 213 | 227
percent change | -0.19 (1.44) | -14.34 (2.06)
Statistical Analysis 1: Comparison: Placebo vs Etelcalcetide; Test type: Superiority or Other; p < 0.001, Repeated Measures Mixed Effects Model; [statistical method as in outcome 3, analysis 1]; Mean Difference = -14.99, 95% CI 2-sided [-19.73 to -10.25], Standard Error of Mean 2.41 — Etelcalcetide - Placebo

6. Secondary Outcome: Percent Change From Baseline in Predialysis Phosphorus During the Efficacy Assessment Phase
Time Frame: Baseline and the efficacy assessment phase (Week 20 to Week 27)
Population: Full analysis set participants with observed data
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Etelcalcetide
Number analyzed (Participants) | 214 | 227
percent change | -1.31 (1.42) | -7.71 (2.16)
Statistical Analysis 1: Comparison: Placebo vs Etelcalcetide; Test type: Superiority or Other; p = 0.003, Repeated Measures Mixed Effects Model; [statistical method as in outcome 3, analysis 1]; Mean Difference = -7.45, 95% CI 2-sided [-12.31 to -2.59], Standard Error of Mean 2.47 — Etelcalcetide - Placebo

ADVERSE EVENTS:
Time Frame: From Day 1 until 30 days after the last dose; the treatment period was 26 weeks.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo | Etelcalcetide
Serious Adverse Events (participants affected / at risk) | 78/254 | 68/251
Other Adverse Events (participants affected / at risk) | 110/254 | 194/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=254) | Etelcalcetide (N=251)
Anaemia (Blood and lymphatic system disorders) | 4 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 6
Angina unstable (Cardiac disorders) | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 4 | 3
Atrial flutter (Cardiac disorders) | 1 | 1
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 1 | 3
Cardiogenic shock (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 2
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 2
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 1 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastrointestinal telangiectasia (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Tooth impacted (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Brain death (General disorders) | 1 | 0
Chills (General disorders) | 2 | 0
Death (General disorders) | 0 | 1
Device issue (General disorders) | 0 | 1
Impaired healing (General disorders) | 1 | 0
Malaise (General disorders) | 2 | 0
Medical device complication (General disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 2 | 3
Pyrexia (General disorders) | 3 | 0
Thrombosis in device (General disorders) | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 1 | 0
Kidney transplant rejection (Immune system disorders) | 1 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Arteriovenous graft site infection (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Diabetic foot infection (Infections and infestations) | 1 | 0
Endocarditis bacterial (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
H1N1 influenza (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 2
Osteomyelitis acute (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 6
Sepsis (Infections and infestations) | 3 | 2
Septic embolus (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Subacute endocarditis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 2
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 3 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Graft haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 1 | 0
Perirenal haematoma (Injury, poisoning and procedural complications) | 1 | 0
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1
Shunt thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0
Anticoagulation drug level above therapeutic (Investigations) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 5 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 4
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Biliary cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bone giant cell tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 2 | 1
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 2 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Accelerated hypertension (Vascular disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1
Blood pressure fluctuation (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Granulomatosis with polyangiitis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Hypertensive emergency (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 2
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 1
Peripheral artery stenosis (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 1
Shock (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
Vascular rupture (Vascular disorders) | 1 | 0
Vascular stenosis (Vascular disorders) | 1 | 0
Venous stenosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=254) | Etelcalcetide (N=251)
Diarrhoea (Gastrointestinal disorders) | 17 | 18
Nausea (Gastrointestinal disorders) | 13 | 31
Vomiting (Gastrointestinal disorders) | 18 | 25
Nasopharyngitis (Infections and infestations) | 13 | 11
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 14 | 11
Blood calcium decreased (Investigations) | 21 | 153
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 18
Muscle spasms (Musculoskeletal and connective tissue disorders) | 18 | 30
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 17
Headache (Nervous system disorders) | 20 | 18
Paraesthesia (Nervous system disorders) | 3 | 13
Hypertension (Vascular disorders) | 16 | 12
Hypotension (Vascular disorders) | 10 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.